CLINICAL TRIAL: NCT04876469
Title: The Role of Radiocontrast Media in Pulsed Radiofrequency Treatment of Lumbar Dorsal Root Ganglion
Brief Title: Radiocontrast Media in the Pulsed Radiofrequency Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Serdar Kokar, Pain Management Physician, M.D., Sanliurfa Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01.02.2021-E.7779
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Lumbar Radiculopathy; Pain, Intractable
Keywords: pulsed radiofrequency treatment; lumbar radicular pain; fluoroscopy
MeSH Terms: conditions — Radiculopathy; Pain, Intractable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiocontrast media group (Active Comparator): Pulsed radiofrequency (PRF) treatment will be applied to the dorsal root ganglion (DRG) by fluoroscopy-guidance at the level of nerve root compression due to disc herniation (L5 level) in both groups.
  In patients in the Radiocontrast media group, contrast material will be given before the application, and primarily the localization of the DRG will be determined. After this stage, the needle will be directed towards the detected localization. Finally, the localization of the dorsal root ganglion will be confirmed by sensory and motor stimuli.
  Interventions: Procedure: Pulsed Radiofrequency treatment of the lumbar dorsal root ganglion
- Non-radiocontrast media group (Active Comparator): Pulsed radiofrequency (PRF) treatment will be applied to the dorsal root ganglion (DRG) by fluoroscopy-guidance at the level of nerve root compression due to disc herniation (L5 level).
  In patients in the Non-radiocontrast media group, the localization of the dorsal root ganglion will be determined just by sensory and motor stimuli.
  Interventions: Procedure: Pulsed Radiofrequency treatment of the lumbar dorsal root ganglion

INTERVENTIONS:
Procedure: Pulsed Radiofrequency treatment of the lumbar dorsal root ganglion — Using radiocontrast media or not for the pulsed radiofrequency treatment of the lumbar dorsal root ganglion

SUMMARY:
Pulsed radiofrequency applied to the dorsal root ganglion (DRG) is an interventional treatment alternative in the treatment of lumbar radicular pain that does not respond to conservative methods. Under intermittent fluoroscopic imaging, the location of the ganglion can be determined by administering contrast media. We consider that determining the localization of the ganglion with this method during pulse radiofrequency application can shorten the procedure time. In this way, we believe that it would help the correct application of the procedure.

DETAILED DESCRIPTION:
Although there are many reasons that can lead to low back pain, radicular pain, which is mostly secondary to lumbar disc hernia, is one of the most common pathologies. Pulsed radiofrequency applied to the dorsal root ganglion (DRG) is an interventional treatment alternative in the treatment of lumbar radicular pain that does not respond to conservative methods and epidural injection treatments.

The electrical field created by the application of pulsed radiofrequency (PRF) changes the cellular activity in DRG neurons. By polarizing cell membranes, reduces nociceptive transmission and contributes to analgesia. In lumbar dorsal root ganglion PRF applications, when the targeted point is reached, the position is confirmed by giving motor and sensory stimuli, and the PRF application is initiated in the follow-up. However, it is a problem that the DRG is not always in the same location, and therefore, time is often lost or even not found while searching with stimulation. Under intermittent fluoroscopic imaging, the location of the ganglion can be determined by administering contrast material.

We consider that determining the localization of the ganglion with this method during pulse radiofrequency application can shorten the procedure time. In this way, we believe that it would help the correct application of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age.
* Lumbar radicular pain
* Lack of response to conservative methods
* L5 nerve root compression due to disc herniation

Exclusion Criteria:

* Patients younger than 18 and older than 65
* Non-radicular low back pain
* L5 nerve root compression due to reasons other than disc herniation
* Those having spondylolisthesis, or transitional vertebra
* Having an active infection
* Pregnancy
* Bleeding diathesis
* Renal Insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Procedure time | 3 months
  The time from cutaneous anesthesia to confirmation of the dorsal root ganglion position by motor and sensory stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moon HS, Kim YD, Song BH, Cha YD, Song JH, Lee MH. Position of dorsal root ganglia in the lumbosacral region in patients with radiculopathy. Korean J Anesthesiol. 2010 Dec;59(6):398-402. doi: 10.4097/kjae.2010.59.6.398. Epub 2010 Dec 31. PMID 21253377
- [Background] Liem L, van Dongen E, Huygen FJ, Staats P, Kramer J. The Dorsal Root Ganglion as a Therapeutic Target for Chronic Pain. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):511-9. doi: 10.1097/AAP.0000000000000408. PMID 27224659
- [Background] Vanneste T, Van Lantschoot A, Van Boxem K, Van Zundert J. Pulsed radiofrequency in chronic pain. Curr Opin Anaesthesiol. 2017 Oct;30(5):577-582. doi: 10.1097/ACO.0000000000000502. PMID 28700369
- [Background] Malik K, Benzon HT. Radiofrequency applications to dorsal root ganglia: a literature review. Anesthesiology. 2008 Sep;109(3):527-42. doi: 10.1097/ALN.0b013e318182c86e. PMID 18719452